CLINICAL TRIAL: NCT02047500
Title: An Open-Label, Phase I Dose Escalation Trial of TH-302 in Combination With Gemcitabine and Nab-Paclitaxel in Previously Untreated Subjects With Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: Phase I TH-302 Plus Gemcitabine Plus Nab-Paclitaxel in Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial has been terminated earlier following the company decision to discontinue the clinical development of Evofosfamide
Sponsor: ImmunoGenesis (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200592-006
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: TH-302; Nab-paclitaxel; Gemcitabine; Evofosfamide
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — TH 302; 130-nm albumin-bound paclitaxel; Gemcitabine

ARMS (1):
- TH-302 plus Nab-paclitaxel plus Gemcitabine (Experimental)
  Interventions: Drug: TH-302; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered at a dose ranging from 170-340 milligram per square meter (mg/m^2) as intravenous infusion over 30 minutes on Days 1, 8 and 15 of every 28-day cycle until evidence of progressive disease, intolerable toxicity or subject withdrawal.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered at a dose ranging from 100-125 mg/m^2 as intravenous infusion over 30 minutes on Days 1, 8 and 15 of every 28-day cycle until evidence of progressive disease, intolerable toxicity or subject withdrawal.
Drug: Gemcitabine — Gemcitabine will be administered at a dose ranging from 800-1000 mg/m^2 as intravenous infusion over 30 minutes on Days 1, 8 and 15 of every 28-day cycle until evidence of progressive disease, intolerable toxicity or subject withdrawal.

SUMMARY:
This is a multicenter, open-label, Phase 1, dose escalation trial to evaluate the safety, tolerability, and recommended Phase 2 dose (RP2D) of TH-302 in combination with gemcitabine and nab-paclitaxel in previously untreated subjects with locally advanced unresectable or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to (>=) 18 years of age with locally advanced unresectable or metastatic pancreatic adenocarcinoma proven by histology or cytology and previously untreated with chemotherapy or systemic therapy other than:

  * Radiosensitizing doses of 5-fluorouracil;
  * Radiosensitizing doses of gemcitabine if relapse occurred at least 6 months after completion of gemcitabine;
  * Neoadjuvant chemotherapy if relapse occurred at least 6 months after surgical resection;
  * Adjuvant chemotherapy if relapse occurred at least 6 months after completion of adjuvant chemotherapy
* Subjects may have measurable or non-measurable disease according to RECIST 1.1.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Acceptable hematological status, liver and renal function as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Significant cardiac or peripheral vascular arterial disease
* Known brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 3 months)
* Severe chronic obstructive or other pulmonary disease with hypoxemia
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Subjects receiving concomitant treatment with radiotherapy or other investigational drugs
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Sun JD, Liu Q, Ahluwalia D, Li W, Meng F, Wang Y, Bhupathi D, Ruprell AS, Hart CP. Efficacy and safety of the hypoxia-activated prodrug TH-302 in combination with gemcitabine and nab-paclitaxel in human tumor xenograft models of pancreatic cancer. Cancer Biol Ther. 2015;16(3):438-49. doi: 10.1080/15384047.2014.1003005. PMID 25679067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TH-302 Plus Nab-paclitaxel Plus Gemcitabine
Started | 19
Completed | 0
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | TH-302 Plus Nab-paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Dose Limiting Toxicity (DLT)
Time Frame: Up to Day 28 of Cycle 1
Population: One patient not evaluable as they did not complete cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | TH-302 Plus Nab-paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Progression Free Survival (PFS) Time
Time Frame: Time from enrollment to progressive disease (PD) or occurrence of death due to any cause within 120 days of either first administration of study drug or the last tumor assessment
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Subjects With Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1) Criteria
Time Frame: Every 8 weeks from Day 1 of Cycle 1 until disease progression or within 1 week after discontinuation of study treatment
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Overall Response According to RECIST Version 1.1 Criteria
Time Frame: Every 8 weeks from Day 1 of Cycle 1 until disease progression or within 1 week after discontinuation of study treatment
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Subjects With Disease Control According to RECIST Version 1.1 Criteria
Time Frame: Every 8 weeks from Day 1 of Cycle 1 until disease progression or within 1 week after discontinuation of study treatment
Reporting Status: Not Posted

6. Secondary Outcome: Tumor Metabolic Response Assessed by Positron Emission Tomography (PET) Scans According to European Organization for Research and Treatment of Cancer (EORTC) Criteria
Time Frame: Baseline and 8 weeks after Day 1 of Cycle 1
Reporting Status: Not Posted

7. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Day 30 after the last dose of study treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | TH-302 Plus Nab-paclitaxel Plus Gemcitabine
Serious Adverse Events (participants affected / at risk) | 19/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 Plus Nab-paclitaxel Plus Gemcitabine (N=19)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 Plus Nab-paclitaxel Plus Gemcitabine (N=19)
Oral herpes (Infections and infestations) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 13 (57)
Leukopenia (Blood and lymphatic system disorders) | 8 (132)
Neutropenia (Blood and lymphatic system disorders) | 14 (88)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (99)
Decreased appetite (Metabolism and nutrition disorders) | 9 (14)
Dehydration (Metabolism and nutrition disorders) | 3 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (21)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Flushing (Vascular disorders) | 3 (6)
Hot flush (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (10)
Abdominal pain lower (Gastrointestinal disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 9 (12)
Flatulence (Gastrointestinal disorders) | 2 (5)
Nausea (Gastrointestinal disorders) | 13 (20)
Proctalgia (Gastrointestinal disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 9 (17)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (15)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 10 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Chills (General disorders) | 8 (13)
Fatigue (General disorders) | 14 (27)
Infusion site rash (General disorders) | 2 (2)
Mucosal inflammation (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 8 (12)
Pyrexia (General disorders) | 7 (12)
Neutrophil count decreased (Investigations) | 3 (11)
Weight decreased (Investigations) | 6 (11)
White blood cell count decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No